CLINICAL TRIAL: NCT03218527
Title: Influence of Circulating Endothelial Progenitor Cells and Modifiable Vascular Risk Factors on Carotid Plaque Vulnerability
Acronym: IMPROVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ATE-2015-38
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Atherosclerosis; Stroke; Inflammation
MeSH Terms: conditions — Atherosclerosis; Stroke; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ischemic stroke is a leading cause of death and disability worldwide. Atherosclerosis, responsible for the 20% of ischemic strokes, is characterized by lipid accumulation in the artery wall that leads to chronic inflammation, cell proliferation and ultimately to vessel stenosis. One of the main features related to plaque progression and vulnerability is inflammation. Positron emission tomography with 18-fluorodeoxyglucos (18-FDG PET) allows an accurate quantification of plaque inflammation and it has been proved its usefulness in predicting early stroke recurrences. The investigators aim to test how modifiable vascular risk factors influence plaque inflammation assessed by 18-FDG PET. In addition, investigators will assess the association of this inflammation and circulating endothelial progenitor cells

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke within 7 days before inclusion
* At least one atherosclerotic plaque in the internal carotid artery
* >18 years old

Exclusion Criteria:

* Cardioembolic strokes according to TOAST criteria
* Poor functional outcome (Rankin >3) after stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed of ischemic stroke presenting at least on atherosclerotic plaque in the internal carotid artery ipsilateral to stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-10-01; Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Standardized Uptake Value (SUV) of the internal carotid artery | Baseline and at one year follow-up
  Inflammation change of the internal carotid artery assessed by the Standardized Uptake Value (SUV) obtained with 18FDG-PET scan at one-year follow-up
Change in the Target-to-Background Ratio (TBR) of the internal carotid artery | Baseline and at one year follow-up
  Inflammation change of the internal carotid artery assessed by the Target-to-Background Ratio (TBR) obtained with 18FDG-PET scan at one-year follow-up
Change in the Endothelial Progenitor Cells Count | Baseline and at one year follow-up
  Change in the Endothelial Progenitor Cells Count by flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia E, Camps-Renom P, Puig N, Fernandez-Leon A, Aguilera-Simon A, Benitez-Amaro A, Sole A, Vilades D, Sanchez-Quesada JL, Marti-Fabregas J, Jimenez-Xarrie E, Benitez S, Llorente-Cortes V. Soluble low-density lipoprotein receptor-related protein 1 as a surrogate marker of carotid plaque inflammation assessed by 18F-FDG PET in patients with a recent ischemic stroke. J Transl Med. 2023 Feb 19;21(1):131. doi: 10.1186/s12967-022-03867-w. PMID 36805772